CLINICAL TRIAL: NCT02952638
Title: Dietary Sources of Lysophospholipids
Status: Terminated | Type: Observational
Sponsor: Susan Smyth (Other)
Responsible Party: Sponsor-Investigator, Susan Smyth, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 14-1001-FIV
Record Dates: First submitted 2015-12-04; First posted 2016-11-02 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Obesity; Cardiovascular Risk Factor; Hyperlipidemia
Keywords: Lipids; lysophosphatidic acid; Lysophospholipids; phosphatidylcholine; lysophosphatidylcholine; autotaxin; dietary
MeSH Terms: conditions — Obesity; Hyperlipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples to measure lysophosphilipid levels
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy: BMI is between 20 and 25
- Overweight: BMI is between 25 and 30
- Obese: BMI is between 30 and 40

SUMMARY:
This study aims to test the hypothesis that dietary intake of phosphatidylcholine (PC) and lysophosphatidylcholine (LPC) acutely alters plasma lysophosphatidic acid (LPA) levels and autotaxin activity in normal weight and obese subjects.

DETAILED DESCRIPTION:
Lysophosphatidic acid (LPA) is a simple glycerophospholipid that is found at biologically-relevant levels in plasma and has important effects on isolated or cultured blood, vascular and fat cells. The main enzyme responsible for generation of plasma LPA is the secreted lysophospholipase D, autotaxin (ATX). Adipocytes contribute substantially to plasma ATX levels. The investigators have demonstrated rapid production and metabolism of plasma LPA in animals. More recently, the investigators have observed that plasma LPA levels increase in mice fed a high fat ("Western") diet in comparison to levels found in mice fed normal chow. The investigators have also found that diet-induced obesity increased circulating ATX levels in mice. The investigators hypothesize that diet, and in particular dietary phosphatidylcholine (PC), may regulate the autotaxin substrate lysophosphatidylcholine (LPC), from which LPA is derived. Obesity may amplify the response by increasing plasma ATX levels and/or activity. The current study will test whether dietary PC in normal weight and obese subjects acutely alters LPA levels and autotaxin activity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years old
* Body Mass Index of 20 and above
* Must be able to consume a low fat meal, unlimited fruits and vegetables and not eating after midnight the night before the lipid tolerance test
* Report to the clinical research unit fasting (no food since the meal the night before)
* Able to consume a liquid meal consisting of a commercial nutritional product supplemented with fat
* Able to have an indwelling catheter placed on one arm and have hourly blood draws for 8 hours

Exclusion Criteria:

* Unstable medical condition (recent or unstable cardiovascular disease)
* Active cancer
* Renal insufficiency Glomerular Filtration Rate <30
* Use of steroids
* Chronic inflammatory conditions
* Use of anticoagulants, anti-inflammatory, or lipid-lowering medications
* Lipodystrophy
* GI conditions that result in lipid intolerance
* Pregnant women have a tendency to be anemic and therefore will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects 18 years of age or older with no major health issues
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-07-14 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Plasma Autotaxin-dependent formation of Lysophosphatidic acid, and Levels of Phosphatidylcholine and its metabolites - Lysophosphatidylcholine, Lysophosphatidic acid, Choline, Trimethylamine and Trimethylamine oxide measured by Tandem Mass Spectrometry | 8 hours
  Investigators will use tandem mass spectrometry to measure the most abundant metabolite species. Enzymatic activity of autotaxin involves incubation with the substrate lysophosphatidylcholine and monitoring concentration dependent release of lysophosphatidic acid. Levels of Lysophospholipids Phosphatidylcholine and the products of its metabolism in the blood will be measured. Quantitation will be achieved by stable isotope dilution and by reference to offline calibration curves. By using mass spectrometry and metabolic tracers, studies using a common protocol are effectively multiplexed so data on both endogenous and mass labeled lipids can be obtained from a single individual. Given the sensitivity of these analytical methods (limits of quantitation of approximately 1 fmol), the measurements and the quantities will be reported as concentration in picomoles per liter of plasma volume. A statistical correlation with each group based on BMI will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Smyth, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Dept of Cardiology, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data.